CLINICAL TRIAL: NCT05335967
Title: Development and Effectiveness Evaluation of a Self-management Program for Prostate Cancer Survivors
Brief Title: Effectiveness Evaluation of a Self-management Program for Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chang Gung Memorial Hospital (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ching-Hui Chien, RN, PhD, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 201902235B0C601
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2023-09

CONDITIONS: Prostatic Neoplasms; Self-Management
Keywords: Prostate cancer; Self-Management; Social participation; Resilience; Rear of cancer recurrence; Self-efficacy; Demoralization
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-management group (Experimental): The experimental group will receive the self-management program for 12 weeks.
  Interventions: Behavioral: Self-management program
- Information group (Other): The control group will receive an information package on a healthy diet.
  Interventions: Other: Information package

INTERVENTIONS:
Behavioral: Self-management program — The self-management group will receive the self-management program for 12 weeks, including a self-management application, a self-management manual, and Professional support.
  Arms: Self-management group
Other: Information package — The patients in this group will receive an information package on a healthy diet.
  Arms: Information group

SUMMARY:
Objectives: This project aims to develop a self-management program for survivors with prostate cancer experiencing urinary incontinence following radical prostatectomy and determine its effectiveness.

Methods: The investigators will develop a self-management program and conduct a study on survivors with prostate cancer experiencing urinary incontinence following radical prostatectomy. And the investigators will test the effectiveness of the self-management program. After completing a pretest, participants will be randomly assigned to the experimental or control group. The self-management group will receive the self-management program for 12 weeks, whereas the information group will receive an information package on a healthy diet. Posttests will be administered 12 and 16 weeks after the pretest. The study variables will include physical symptoms and bothers, cancer-related self-efficacy, social participation, demoralization, and resilience.

DETAILED DESCRIPTION:
Objectives: This project aims to develop a self-management program for survivors with prostate cancer experiencing urinary incontinence following radical prostatectomy and determine its effectiveness.

Methods: The investigators will develop a self-management program and conduct a study on survivors with prostate cancer experiencing urinary incontinence following radical prostatectomy. And the investigators will test the effectiveness of the self-management program. After completing a pretest, participants will be randomly assigned to the experimental or control group. The self-management group will receive the self-management program for 12 weeks, whereas the information group will receive an information package on a healthy diet. The self-management program is included a self-management application, a self-management manual, and professional support. The information package consists of a manual on a healthy diet and a multimedia film on a healthy diet. Posttests will be administered 12 and 16 weeks after the pretest. The study variables will include physical symptoms and bothers, cancer-related self-efficacy, social participation, demoralization, and resilience. The statistical analyses will consist of independent sample t-tests, Chi-squire, and generalized estimating equation analysis.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer survivors will include if they fit the following:

* Received radical prostatectomy and suffering from urinary incontinence for at least one week
* Eastern Cooperative Oncology Group 0-1 point, able to walk entirely independently
* Have a smartphone or a tablet with a wireless network
* Their intimate partner or one of the family members willing to learn together
* Agreed to participate in the study and completed the informed consent form

Exclusion Criteria:

Prostate cancer survivors will be excluded if they had one or more of the following:

* A request, with the consideration of family members, that the medical team not tell the patient about the diagnosis or condition of the disease
* A history of psychiatric illness, such as dementia, depression; schizophrenia, or bipolar disorder
* Suffer from other types of cancer and actively undergoing treatment

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Cancer related self-efficacy | Pre-test
  The Mandarin version of the Cancer Survivors' Self-Efficacy Scale (CSSES) will be used to evaluate the cancer-specific self-efficacy of participants.The total score ranges from 11 to 110; the lower the score, the worse the self-efficacy.
Cancer related self-efficacy | 12 weeks after the pretest
  The Mandarin version of the Cancer Survivors' Self-Efficacy Scale (CSSES) will be used to evaluate the cancer-specific self-efficacy of participants.The total score ranges from 11 to 110; the lower the score, the worse the self-efficacy.
Cancer related self-efficacy | 16 weeks after the pretest
  The Mandarin version of the Cancer Survivors' Self-Efficacy Scale (CSSES) will be used to evaluate the cancer-specific self-efficacy of participants.The total score ranges from 11 to 110; the lower the score, the worse the self-efficacy.

SECONDARY OUTCOMES:
Urinary symptoms and bothers | Pre-test
  The Mandarin version of the Expanded Prostate Cancer Index Composite (EPIC) will be used to measure the urinary symptoms and bother of the participants. Total 7 items and each question is linearly scaled from 0 (worst) to 100 (best).
Urinary symptoms and bothers | 12 weeks after the pretest
  The Mandarin version of the Expanded Prostate Cancer Index Composite (EPIC) will be used to measure the urinary symptoms and bother of the participants. Total 7 items and each question is linearly scaled from 0 (worst) to 100 (best).
Urinary symptoms and bothers | 16 weeks after the pretest
  The Mandarin version of the Expanded Prostate Cancer Index Composite (EPIC) will be used to measure the urinary symptoms and bother of the participants. Total 7 items and each question is linearly scaled from 0 (worst) to 100 (best).
Social participation | Pre-test
  A. The Mandarin version of the Older Adults Social Participation Scale will be used to assess participants' social participation. The scale includes 12 items with a score range of 12 to 60. A higher score shows a higher degree of social participation.
  B. Self-designed items will be used to assess participants' willingness to participate in social activities (1 item) and their satisfaction with social activities (1 item). Each item will have a score range of 0 to 10, with higher scores indicating a greater willingness to participate or higher satisfaction.
Social participation | 12 weeks after the pretest
  A. The Mandarin version of the Older Adults Social Participation Scale will be used to assess participants' social participation. The scale includes 12 items with a score range of 12 to 60. A higher score shows a higher degree of social participation.
  B. Self-designed items will be used to assess participants' willingness to participate in social activities (1 item) and their satisfaction with social activities (1 item). Each item will have a score range of 0 to 10, with higher scores indicating a greater willingness to participate or higher satisfaction.
Social participation | 16 weeks after the pretest
  A. The Mandarin version of the Older Adults Social Participation Scale will be used to assess participants' social participation. The scale includes 12 items with a score range of 12 to 60. A higher score shows a higher degree of social participation.
  B. Self-designed items will be used to assess participants' willingness to participate in social activities (1 item) and their satisfaction with social activities (1 item). Each item will have a score range of 0 to 10, with higher scores indicating a greater willingness to participate or higher satisfaction.
Demoralization | Pre-test
  The Mandarin version of the Demoralization Scale will be used to assess participants' demoralization. The scale includes 24 items, and the score range is 0-96. A higher score means higher demoralization.
Demoralization | 12 weeks after the pretest
  The Mandarin version of the Demoralization Scale will be used to assess participants' demoralization. The scale includes 24 items, and the score range is 0-96. A higher score means higher demoralization.
Demoralization | 16 weeks after the pretest
  The Mandarin version of the Demoralization Scale will be used to assess participants' demoralization. The scale includes 24 items, and the score range is 0-96. A higher score means higher demoralization.
Resilience | Pre-test
  The Mandarin version of the Connor-Davidson Resilience Scale will be used to measure the psychological resilience of participants. The scale has 10 items, and the score range is 0-100. A higher score reflects better resilience.
Resilience | 12 weeks after the pretest
  The Mandarin version of the Connor-Davidson Resilience Scale will be used to measure the psychological resilience of participants. The scale has 10 items, and the score range is 0-100. A higher score reflects better resilience.
Resilience | 16 weeks after the pretest
  The Mandarin version of the Connor-Davidson Resilience Scale will be used to measure the psychological resilience of participants. The scale has 10 items, and the score range is 0-100. A higher score reflects better resilience.

OTHER OUTCOMES:
Demographic characteristic and disease information list 1 | Pre-test
  Age
Demographic characteristic and disease information list 2 | Pre-test
  Marital status
Demographic characteristic and disease information list 3 | Pre-test
  Education level
Demographic characteristic and disease information list 4 | Pre-test
  Religious beliefs
Demographic characteristic and disease information list 5 | Pre-test
  Employment status
Demographic characteristic and disease information list 6 | Pre-test
  Cancer stage
Demographic characteristic and disease information list 7 | Pre-test
  Chronic disease history
Demographic characteristic and disease information list 8 | Pre-test
  Time of diagnosis (months)
Demographic characteristic and disease information list 9 | Pre-test
  Treatment methods
Demographic characteristic and disease information list 10 | Pre-test
  Latest serum level of prostate-specific antigen (ng/mL)
Demographic characteristic and disease information list 11 | 12 weeks after the pretest
  Latest serum level of prostate-specific antigen (ng/mL)
Demographic characteristic and disease information list 12 | 16 weeks after the pretest
  Latest serum level of prostate-specific antigen (ng/mL)
Satisfaction and evaluation of self-management intervention | 12 weeks after the pretest
  Self-designed five items will be used to assess these outcomes.Each item is scaled from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hui Chien, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences, Taipei, Taiwan.
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital at Keelung, Keelung
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien CH, Liu KL, Wu CT, Chuang CK, Yu KJ, Lin PH, Huang XY, Pang ST. Development and assessment of a self-management intervention for urinary incontinence among patients with prostate cancer: protocol for a randomized feasibility study. BMC Urol. 2023 Nov 18;23(1):193. doi: 10.1186/s12894-023-01367-7. PMID 37980490
- [Background] Agochukwu NQ, Skolarus TA, Wittmann D. Telemedicine and prostate cancer survivorship: a narrative review. Mhealth. 2018 Oct 8;4:45. doi: 10.21037/mhealth.2018.09.08. eCollection 2018. PMID 30505843
- [Background] An E, Lo C, Hales S, Zimmermann C, Rodin G. Demoralization and death anxiety in advanced cancer. Psychooncology. 2018 Nov;27(11):2566-2572. doi: 10.1002/pon.4843. Epub 2018 Aug 20. PMID 30053317
- [Background] Baker H, Wellman S, Lavender V. Functional Quality-of-Life Outcomes Reported by Men Treated for Localized Prostate Cancer: A Systematic Literature Review. Oncol Nurs Forum. 2016 Mar;43(2):199-218. doi: 10.1188/16.ONF.199-218. PMID 26906131
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Chien CH, Chuang CK, Liu KL, Huang XY, Liu HE. Psychosocial adjustments in patients with prostate cancer from pre-diagnosis to 6 months post-treatment. Int J Nurs Pract. 2016 Feb;22(1):70-8. doi: 10.1111/ijn.12360. Epub 2014 Oct 13. PMID 25307968
- [Background] Chien CH, Chung HJ, Liu KL, Pang ST, Wu CT, Chang YH, Huang XY, Chang YH, Lin TP, Lin WY, Chuang CK. Effectiveness of a couple-based psychosocial intervention on patients with prostate cancer and their partners: A quasi-experimental study. J Adv Nurs. 2020 Oct;76(10):2572-2585. doi: 10.1111/jan.14471. Epub 2020 Aug 3. PMID 32744426
- [Background] Chou MC, Chien CH, Chung HJ, Chuang CK, Wu CT, Pang ST, Liu KL, Chang YH. The Psychometric Properties of Taiwanese Version of the Memorial Anxiety Scale for Prostate Cancer. J Pain Symptom Manage. 2021 Apr;61(4):824-830. doi: 10.1016/j.jpainsymman.2020.10.013. Epub 2020 Oct 24. PMID 33198956
- [Background] Cockle-Hearne J, Faithfull S. Self-management for men surviving prostate cancer: a review of behavioural and psychosocial interventions to understand what strategies can work, for whom and in what circumstances. Psychooncology. 2010 Sep;19(9):909-22. doi: 10.1002/pon.1657. PMID 20119934
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Crafoord MT, Fjell M, Sundberg K, Nilsson M, Langius-Eklof A. Engagement in an Interactive App for Symptom Self-Management during Treatment in Patients With Breast or Prostate Cancer: Mixed Methods Study. J Med Internet Res. 2020 Aug 10;22(8):e17058. doi: 10.2196/17058. PMID 32663140
- [Background] Faithfull S, Cockle-Hearne J, Khoo V. Self-management after prostate cancer treatment: evaluating the feasibility of providing a cognitive and behavioural programme for lower urinary tract symptoms. BJU Int. 2011 Mar;107(5):783-790. doi: 10.1111/j.1464-410X.2010.09588.x. Epub 2010 Oct 13. PMID 20942826
- [Background] Foster C, Breckons M, Cotterell P, Barbosa D, Calman L, Corner J, Fenlon D, Foster R, Grimmett C, Richardson A, Smith PW. Cancer survivors' self-efficacy to self-manage in the year following primary treatment. J Cancer Surviv. 2015 Mar;9(1):11-9. doi: 10.1007/s11764-014-0384-0. Epub 2014 Jul 16. PMID 25028218
- [Background] Foster C, Fenlon D. Recovery and self-management support following primary cancer treatment. Br J Cancer. 2011 Nov 8;105 Suppl 1(Suppl 1):S21-8. doi: 10.1038/bjc.2011.419. PMID 22048029
- [Background] Frankland J, Brodie H, Cooke D, Foster C, Foster R, Gage H, Jordan J, Mesa-Eguiagaray I, Pickering R, Richardson A. Follow-up care after treatment for prostate cancer: evaluation of a supported self-management and remote surveillance programme. BMC Cancer. 2019 Apr 23;19(1):368. doi: 10.1186/s12885-019-5561-0. PMID 31014282
- [Background] Jonkman NH, Schuurmans MJ, Groenwold RHH, Hoes AW, Trappenburg JCA. Identifying components of self-management interventions that improve health-related quality of life in chronically ill patients: Systematic review and meta-regression analysis. Patient Educ Couns. 2016 Jul;99(7):1087-1098. doi: 10.1016/j.pec.2016.01.022. Epub 2016 Feb 1. PMID 26856778
- [Background] Kissane DW, Wein S, Love A, Lee XQ, Kee PL, Clarke DM. The Demoralization Scale: a report of its development and preliminary validation. J Palliat Care. 2004 Winter;20(4):269-76. PMID 15690829
- [Background] Xu A, Wang Y, Wu X. Effectiveness of e-health based self-management to improve cancer-related fatigue, self-efficacy and quality of life in cancer patients: Systematic review and meta-analysis. J Adv Nurs. 2019 Dec;75(12):3434-3447. doi: 10.1111/jan.14197. Epub 2019 Oct 20. PMID 31566769
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Straczynska A, Weber-Rajek M, Strojek K, Piekorz Z, Styczynska H, Goch A, Radziminska A. The Impact Of Pelvic Floor Muscle Training On Urinary Incontinence In Men After Radical Prostatectomy (RP) - A Systematic Review. Clin Interv Aging. 2019 Nov 12;14:1997-2005. doi: 10.2147/CIA.S228222. eCollection 2019. PMID 31814714
- [Background] Song L, Guo P, Tan X, Chen RC, Nielsen ME, Birken SA, Koontz BF, Northouse LL, Mayer DK. Enhancing survivorship care planning for patients with localized prostate cancer using a couple-focused web-based, mHealth program: the results of a pilot feasibility study. J Cancer Surviv. 2021 Feb;15(1):99-108. doi: 10.1007/s11764-020-00914-7. Epub 2020 Jul 17. PMID 32681304
- [Background] Skolarus TA, Metreger T, Wittmann D, Hwang S, Kim HM, Grubb RL 3rd, Gingrich JR, Zhu H, Piette JD, Hawley ST. Self-Management in Long-Term Prostate Cancer Survivors: A Randomized, Controlled Trial. J Clin Oncol. 2019 May 20;37(15):1326-1335. doi: 10.1200/JCO.18.01770. Epub 2019 Mar 29. PMID 30925126
- [Background] Sharpley CF, Bitsika V, Christie DRH, Bradford R, Steigler A, Denham JW. Psychological resilience aspects that mediate the depressive effects of urinary incontinence in prostate cancer survivors 10 years after treatment with radiation and hormone ablation. J Psychosoc Oncol. 2017 Jul-Aug;35(4):438-450. doi: 10.1080/07347332.2017.1306733. Epub 2017 Mar 20. PMID 28318448
- [Background] Roth AJ, Rosenfeld B, Kornblith AB, Gibson C, Scher HI, Curley-Smart T, Holland JC, Breitbart W. The memorial anxiety scale for prostate cancer: validation of a new scale to measure anxiety in men with with prostate cancer. Cancer. 2003 Jun 1;97(11):2910-8. doi: 10.1002/cncr.11386. PMID 12767107
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348